CLINICAL TRIAL: NCT06613139
Title: An Open-label, Randomized, Single-dose, Oral Administration, 2-sequence, 2- Period, Crossover Study to Evaluate Bioequivalence Between YHP2305 and YHR2404 in Healthy Subjects
Brief Title: Bioequivalence Study Between YHP2305 and YHR2404 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHP2305-101
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Bioequivalence

STUDY DESIGN:
Intervention Model Description: Crossover Assignment two-way crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A(RT) (Experimental): 17 subjects, Cross-over, Single dose of YHR2404 on day 1, Single dose of YHP2305 on day 8
  Interventions: Drug: YHP2305; Drug: YHR2404
- Group B(TR) (Experimental): 17 subjects, Cross-over, Single dose of YHP2305 on day 1, Single dose of YHR2404 on day 8
  Interventions: Drug: YHP2305; Drug: YHR2404

INTERVENTIONS:
Drug: YHP2305 — Test drug: YHP2305 Comparator: YHR2404
Drug: YHR2404 — Test drug: YHP2305 comparator: YHR2404

SUMMARY:
An open-label, randomized, single-dose, oral administration, 2-sequence, 2- period, crossover study to evaluate bioequivalence between YHP2305 and YHR2404 in healthy subjects

DETAILED DESCRIPTION:
Subjects in group A will be administered comparator and YHP2305 by crossover design on day 1, 8.

Subjects in group B will be administered YHP2305 and comparator by crossover design on day 1, 8.

ELIGIBILITY:
Inclusion Criteria:

* Those who are 19 years old or older at the screening visit
* Those whose weight is over 50kg(male), over 45kg(female) and their body mass index (BMI) shall be between 18.0 kg/m2 and 30.0 kg/m2
* Those who express their voluntary consent to participate in the trial by signing a written consent
* Those who are judged eligible to participate in the trial by the principal investigator(or delegated investigators) after screening test

Exclusion Criteria:

* Those who have participated in a bioequivalence study or other clinical trials and have been administered with investigational products in 6 months prior to the first administration.
* Others who are judged ineligible to participate in the trial by the principal investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-10-06 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve [AUCt] | 0-36 hours
Maximum plasma concentration [Cmax] | 0-36 hours

SECONDARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity [AUCinf] | 0-36 hours
Area under the plasma drug concentration-time curve/Area under the plasma drug concentration-time curve from time 0 to infinity [AUCt/AUCinf] | 0-36 hours
Time of peak concentration [Tmax] | 0-36 hours
Terminal phase of half-life [t1/2] | 0-36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Taegon Hong, Principal Investigator — Locations
Locations (1):
- Bumin Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No